CLINICAL TRIAL: NCT03234387
Title: A CFit Study: To What Extent Does Inflammation, Oxidative Stress, Nitric Oxide Bioavailability and Microvascular Endothelial Dysfunction Influence the Aerobic Exercise Function of Individuals With Cystic Fibrosis, With and Without Established Diabetes?
Brief Title: A CFit Study - Baseline
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: University of Portsmouth (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Loughborough University (Other); Queen Alexandra Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Other Study IDs: ZS002
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis-related Diabetes
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise Test; Insulin; Glucose Tolerance Test; Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Acellular plasma will be stored at - 80 degrees
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cystic fibrosis (CF) with established CF-related diabetes: Cystic fibrosis (CF) with established CF-related diabetes
  Inclusion criteria:
  * Males and females ≥ 12 years of age
  * CF diagnosis based on clinical features, supported by an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat) and, where possible, diagnostic genotyping
  * Established CFRD in accordance with the most recent American Diabetes Association positional statement]. This statement recommends CFRD is diagnosed using a 2 hour OGTT. However, the present study will also include those based on fasting plasma glucose and glycated hemoglobin levels, when symptoms of diabetes are also present:
    * 2 hour OGTT plasma glucose ≥ 200 mg.dL-1 (11.1 mmol.L-1)
    * Fasting plasma glucose ≥ 126 mg.dL-1 (7.0 mmol.L-1)
    * Glycated hemoglobin ≥ 48 mmol/mol
  * No contraindications to performing exhaustive exercise
  * Can understand and cooperate with the study protocol
  * No increase in symptoms or weight loss in the preceding 2 weeks
  Interventions: Other: No intervention - only assessments.
- Cystic fibrosis (CF) without established CF-related diabetes: Cystic fibrosis (CF) without established CF-related diabetes
  Inclusion criteria:
  * Males and females ≥ 12 years of age
  * CF diagnosis based on clinical features, supported by an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat), where possible, diagnostic genotyping would also be desired
  * No evidence of established, gestational or exacerbation induced CFRD in accordance with the American Diabetes Association criteria (stated above; [110]).
  * No contraindications to performing exhaustive exercise
  * Can understand and cooperate with the study protocol
  * No increase in symptoms or weight loss in the preceding 2 weeks
  Interventions: Other: No intervention - only assessments.
- Healthy controls: Age- and gender-matched healthy control participants.
  Interventions: Other: No intervention - only assessments.

INTERVENTIONS:
Other: No intervention - only assessments. — No intervention only a number of assessments. Participants will be assessed during a maximal cardiopulmonary exercise testing on an exercise bike during 1 visit, and before and after an oral glucose tolerance test on a following visit.
  Other Names: Exercise testing; Insulin and acetylcholine iontophoresis measures of microvascular function; Oral glucose tolerance test (75 g glucose)

SUMMARY:
A great medical success is the increase in the median survival age associated with cystic fibrosis (CF). However, this success has led to a new era of research with the aim to maximise the quality of life (QoL) of the aging CF population. Recent research has demonstrated that the traditional method of determining disease progression, i.e. pulmonary function, no longer adequately predict survival rates. Therefore, various bodies have promoted cardiopulmonary exercise testing (CPET), as outcomes from this test (e.g. one's maximal O2 uptake [VO₂max]) are known predictors of the QoL, risk of hospitalisation and prognosis of individuals with CF.

One of the most common non-pulmonary co-morbidities of CF is CF-related diabetes (CFRD). Importantly, CFRD is associated with a poorer pulmonary function compared to CF patients without CFRD, and ultimately a worsened prognosis. Despite this, the influence an impaired glycaemic control has upon the VO₂max derived from a CPET is unknown in CF. Therefore, the present study aims to assess whether VO₂max, an established determinant of QoL, differs between patients with CF with and without established CFRD as well as a group of age- and gender-matched healthy control subjects.

The additional measures within the present study, such as: biomarkers of inflammation, redox balance and nitric oxide (NO2) bioavailability, as well as functional measures of microvascular endothelial function will aid our knowledge of the physiological abnormalities which are a cause or consequence of CFRD. Importantly, by identifying the factors which may contribute to CFRD progression and those that are viable for early intervention, mean the aims and objectives of this study are compatible with the top 10 research objectives set by the CF Trust.

DETAILED DESCRIPTION:
Participants and recruitment The present study will be a pilot, cross-sectional trial in individuals with CFRD (n = 15), as well as age- and gender-matched CF controls without diabetes (n = 15) and age- and gender-matched healthy control participants (n = 15). Participants will be recruited from adult and paediatric CF outpatient clinics within the Southampton CF network. The healthy control participants will be recruited from the University of Portsmouth and local area. Individuals with CF will be tested at a laboratory established within the CF unit at the Southampton General Hospital and/or the Department of Sport and Exercise Sciences (University of Portsmouth), depending on participant convenience. All healthy control participants will attend the Department of Sport and Exercise Sciences at the University of Portsmouth.

Visit 1 During this visit, a valid informed consent and GCP trained member of the research team will fully explain the information sheet and study protocol, as well as answer any questions to ensure that all relevant parties are clear about the study requirements. Following this, fully informed written consent will be obtained. Additionally, informed written assent will be obtained from those < 16 years of age.

Following the consent procedures the participants resting pulmonary function (forced vital capacity, forced expiratory volume in 1 second, mid force expiratory flow and peak expiratory flow) and anthropometric measures (weight, height and body fat percentage) will obtained. The subsequent aim of this visit is then to habituate all participants with exercising on a cycle ergometer in preparation for their CPET in visit 2, in particular maintaining a certain cadence at a given power output. Appropriate adjustments will be made to the ergometer seat and handlebar position, and noted for visit 2. Furthermore, the protocols of obtaining ones ratings of perceived exertion and dyspnoea will be fully explained. Lastly, the participant will be instructed to avoid consuming mouthwash for the entirety of the study period due to evidence suggesting it may influence the uptake of dietary nitrate.

Visit 2 Participants will arrive to the laboratory at 1900 ± 2 hours. They will be instructed to arrive 2 hours postprandial, having avoided caffeine for > 12 hours, as well as nitrate rich foods, alcohol and exhaustive exercise for > 24 hours.

Upon arrival, CGM's will be fixed to the interior surface of the upper arm and worn for the subsequent 14 days. In addition to this, hip worn accelerometers, as well as hourly specific physical activity and food diaries will be distributed and completed for 14 days alongside the CGM. The participants resting pulmonary function will be assessed using the spirometry procedures described below, and a resting blood sample will be collected via venepuncture for the analysis of plasma [NO-(₂)] and ET-1. Additionally, the cycle ergometer CPET with a supramaximal (Smax) verification phase will be employed to determine ones aerobic exercise function, and a second venous blood sample will be collected immediately following exercise termination for the analysis of plasma [NO-(₂)] and ET-1. The total volume of blood collected over this 2 hour visit will be approximately 20 mL.

Visit 3 Participants will be required to arrive to the laboratory ≥ 3 days post visit 1, at 0800 ± 2 hours, following an overnight fast (> 10 hours). Furthermore, participants will be instructed to avoid nitrate rich foods, caffeine, alcohol and exhaustive exercise for 24 hours prior to arrival.

Upon arrival participants will undergo the acetylcholine (ACh) and insulin iontophoresis protocols described below, including 5 resting blood pressure measurements. Immediately following this, the participant's pulmonary function will be assessed via spirometry. Participants will be asked to rest, and entertainment will be provided, for the following 60 minutes. The iontophoresis procedures will then be repeated to assess the short-term test-retest variability of the iontophoresis procedures. Following this, a cannula will be inserted into a vein by a trained phlebotomist, prior to the 3 hour OGTT and a baseline blood sample will be taken (measuring all the below biomarkers). Venous blood samples will be drawn at 30, 60, 90, 120 and 180 minutes post glucose ingestion for the analysis of glucose, insulin, active glucagon-like peptide-1 (GLP-1), TNF-α, soluble vascular cell adhesion molecule-1 (sVCAM-1), IL-6, [NO-(₂)] and ET-1. NT, total glutathione (tGSH) and total cysteine (tCys) will be analysed at 120 minutes post-glucose ingestion. The total volume of blood collected over this 5 hour visit will be approximately 176 mL. Additionally, the iontophoresis procedures will be repeated at 30, 90 and 150 minutes post-glucose ingestion (i.e. hourly measurements of microvascular endothelial function).

Follow-up CGM's, accelerometers and physical activity/food diaries will be completed for 14 days following visit 1. A member of the research team will collect these from the preferred location of the participant.

ELIGIBILITY:
GROUP 1:

Cystic fibrosis (CF) with established CF-related diabetes:

Inclusion Criteria:

* Males and females ≥ 12 years of age
* CF diagnosis based on clinical features, supported by an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat) and, where possible, diagnostic genotyping
* Established CFRD in accordance with the most recent American Diabetes Association positional statement. This statement recommends CFRD is diagnosed using a 2 hour OGTT. However, the present study will also include those based on fasting plasma glucose and glycated hemoglobin levels, when symptoms of diabetes are also present:

  * 2 hour OGTT plasma glucose ≥ 200 mg.dL-1 (11.1 mmol.L-1)
  * Fasting plasma glucose ≥ 126 mg.dL-1 (7.0 mmol.L-1)
  * Glycated hemoglobin ≥ 48 mmol/mol
* No contraindications to performing exhaustive exercise
* Can understand and cooperate with the study protocol
* No increase in symptoms or weight loss in the preceding 2 weeks

Exclusion Criteria:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (arthritis, joint or muscle disease) and cardiovascular disease (congenital heart disease or cardiomyopathy).
* Unstable co-morbid asthma (daily pulmonary function variability of >20%)
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not of a suitable age for testing

GROUP 2:

Cystic fibrosis (CF) without established CF-related diabetes:

Inclusion Criteria:

* Males and females ≥ 12 years of age
* CF diagnosis based on clinical features, supported by an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat), where possible, diagnostic genotyping would also be desired
* No evidence of established, gestational or exacerbation induced CFRD in accordance with the American Diabetes Association criteria (stated above).
* No contraindications to performing exhaustive exercise
* Can understand and cooperate with the study protocol
* No increase in symptoms or weight loss in the preceding 2 weeks

Exclusion Criteria:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (arthritis, joint or muscle disease) and cardiovascular disease (congenital heart disease or cardiomyopathy).
* Unstable co-morbid asthma (daily pulmonary function variability of >20%)
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not of a suitable age for testing
* Not a suitable age- and gender-match for those with CFRD

Exclusion during testing:

* Onset of acute infection
* Becomes and/or is tested to be pregnant following enrolment to the study
* Unable to understand or cooperate with study protocol
* The individual does not wish to participate further

GROUP 3:

Healthy age- and gender-matched control participants:

Inclusion Criteria:

* Age- and gender

Exclusion Criteria:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (arthritis, joint or muscle disease), respiratory and cardiovascular disease (congenital heart disease or cardiomyopathy).
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not a suitable age- and gender-match for those with CFRD

Exclusion during testing:

* Onset of acute illness or injury
* Becomes and/or is tested to be pregnant following enrolment to the study
* Unable to understand or cooperate with study protocol
* The individual does not wish to participate further

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Individuals with cystic fibrosis (CF) and established CF-related diabetes (CFRD)
  * Individuals with CF and no established CFRD (age- and gender-matched to CFRD group)
  * Healthy age- and gender-matched control participants (matched to CFRD group)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (aerobic fitness) | Visit 1 - Baseline
  Maximal oxygen uptake (aerobic fitness) from a maximal cardiopulmonary exercise testing on a cycle ergometer

SECONDARY OUTCOMES:
VO2 gain | Visit 1 - Baseline
  Oxygen cost of exercise (efficiency) - derived from maximal cardiopulmonary exercise test on a cycle ergometer
VO2 mean response time | Visit 1 - Baseline
  VO2 mean response time - derived from maximal cardiopulmonary exercise test
Gas exchange threshold | Visit 1 - Baseline
  Gas exchange threshold - derived from maximal cardiopulmonary exercise test
Near-infrared spectroscopy derived deoxygenated [haemoglobin + myoglobin] | Visit 1 - Baseline
  Dynamics of near-infrared spectroscopy derived deoxygenated [haemoglobin + myoglobin]
Pulmonary function | Visit 1 (baseline), Visit 2 (baseline)
  Pulmonary function measured using flow-volume loop spirometry
Glycaemic control | Glycaemic control will be measured continuously for 14 days following visit 1.
  Glycaemic control measured using an arm-mounted continuous glucose monitor
Physical activity | Physical activity will be measured continuously for 14 days following visit 1.
  Physical activity measured using a wrist-mounted physical activity monitor
Dietary intake | Food diaries will be completed for 14 days following visit 1.
  Dietary intake measured using MyFitness Pal application and food diaries
Tumour necrosis factor alpha (TNF-alpha) | Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Tumour necrosis factor alpha (TNF-alpha) measured from plasma
Soluble vascular cell adhesion molecule-1 (sVCAM) | Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Soluble vascular cell adhesion molecule-1 (sVCAM) measured from plasma
Endothelin-1 (ET-1) | Visit 1 (baseline and following maximal cardiopulmonary exercise test on cycle ergometer), Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Endothelin-1 (ET-1) measured from plasma
Interleukin-6 (IL-6) | Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Interleukin-6 (IL-6) measured from plasma
[Nitrite] (NO2) | Visit 1 (baseline ), Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Nitrite concentration measured from plasma
Nitrotyrosine (NT) | Visit 2: (baseline) and 120 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Nitrotyrosine (NT) measured from plasma
Total glutathione (tGSH) | Visit 2: (baseline) and 120 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Total glutathione (tGSH) measured from plasma
Total cysteine (tCys) | Visit 2: (baseline) and 120 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Total cysteine (tCys) measured from plasma
Acetylcholine (Ach) iontophoresis | Visit 2: (baseline) and 1, 2 and 3 hours following ingestion of 75 g glucose for an oral glucose tolerance test
  Acetylcholine (Ach) iontophoresis measure of microvascular function
Insulin iontophoresis | Visit 2: (baseline) and 1, 2 and 3 hours following ingestion of 75 g glucose for an oral glucose tolerance
  Insulin iontophoresis measure of microvascular function
Glucose concentration | Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Glucose concentration
Insulin concentration | Visit 2: (baseline) and 30, 60, 90, 120 and 180 minutes following ingestion of 75 g glucose for an oral glucose tolerance test
  Insulin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the study team only.